CLINICAL TRIAL: NCT03941782
Title: INST UNM 1601: Compassionate Use of BYL 719 Alpelisib
Brief Title: Compassionate Use of BYL 719 Alpelisib
Status: No longer available | Type: Expanded Access
Sponsor: New Mexico Cancer Research Alliance (Other)
Responsible Party: Sponsor
Other Study IDs: INST UNM 1601
Record Dates: First submitted 2019-05-06; First posted 2019-05-08 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Lymphangioma
MeSH Terms: conditions — Lymphangioma | interventions — Alpelisib

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Alpelisib — As a single agent, alpelisib will be administered at a starting dose of 350 mg orally once daily on a continuous dosing schedule and can be adjusted for toxicity per the recommendations in this protocol. No pretreatment will be given prior to the medication.
  Other Names: BYL719

SUMMARY:
This is a compassionate use protocol of BYL719 (alpelisib) treatment for a single patient with locally advanced lymphangioma positive PI3K alpha H1047R mutation.

DETAILED DESCRIPTION:
As a single agent, alpelisib will be administered at a starting dose of 350 mg orally once daily on a continuous dosing schedule and can be adjusted for toxicity per the recommendations in this protocol. No pretreatment will be given prior to the medication.

We plan on treating this individual patient for a tentative period of 12 weeks at which time treating physician will reevaluate the patient's clinical and radiological response and further duration of treatment will be contingent on that assessment.

ELIGIBILITY:
Inclusion Criteria:

* Patient eligible for inclusion in this Treatment Plan have to meet all of the following criteria:

  1. Patient has signed the Informed Consent (ICF) prior to any eligibility evaluations being performed and is able to comply with protocol requirements
  2. Patient is an adult and ≥ 18 years old at the time of informed consent
  3. Patient has locally advanced or metastatic cancer resistant or refractory to available standard of care treatment options and has no other available comparable or satisfactory alternative treatment options
  4. PIK3CA mutation, or other molecular alteration known to activate PI3K, in tumor tissue as determined by a standard Laboratory
  5. Patient is not eligible for participation in any ongoing clinical trials with alpelisib, or has recently completed a clinical trial with alpelisib that has been terminated, and after considering other options (e.g. trial extensions, amendments, etc.), the treating physician has determined that treatment is necessary and there are no other feasible alternatives for the patient
  6. Patient is not being transferred from an ongoing clinical trial for which they are still eligible
  7. Patient has adequate bone marrow and organ function as defined by the following laboratory values:

     1. Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L
     2. Platelets ≥ 100 x 109/L (For patients with hematologic malignancies involving the bone marrow, platelet count > 75 x 109/L may be acceptable)
     3. Hemoglobin ≥ 9.0 g/dL
     4. INR ≤ 1.5
     5. Potassium, magnesium and calcium (corrected for albumin), within normal limits for the institution, or ≤ Grade 1 severity according to NCI-CTCAE version 4.03 if judged clinically not significant by the investigator
     6. Serum creatinine ≤ 1.5 x ULN and/or creatinine clearance > 50% LLN (Lower Limit of Normal)
     7. Total serum bilirubin < ULN (or ≤ 1.5 x ULN if liver metastases are present; or total bilirubin ≤ 3.0 x ULN with direct bilirubin within normal range in patients with well documented Gilbert's Syndrome, (defined as presence of several episodes of unconjugated hyperbilirubinemia with normal CBC results including normal reticulocyte count and peripheral blood smear, normal liver function test results, and absence of other contributing disease processes at the time of diagnosis)
     8. Alanine aminotransferase (AST) and aspartate aminotransferase (ALT) ≤ 2.5 ULN (or < 5.0 x ULN if liver metastases are present)
  8. Patient is deemed by the Treating Physician to have the initiative and means to be compliant with the treatment plan (treatment and follow-up requested by the Treating Physician)

Exclusion Criteria:

* Patients eligible for this Treatment Plan must not meet any of the following criteria:

  1. Patient has history of hypersensitivity to any drugs or metabolites of similar chemical classes as alpelisib
  2. Patient has not recovered to grade 1 or better (except alopecia) from related side effects of any prior antineoplastic therapy
  3. Patient has had major surgery within 4 weks prior to starting treatment with alpelisib or has not recovered from major side effects
  4. Patient is currently receiving or has received systemic corticosteroids ≤ 2 weeks prior to starting treatment with alpelisib, or has not fully recovered from side effects of such treatment
  5. Patient with clinically manifest diabetes mellitus, or documented steroid induced diabetes mellitus
  6. Patient is being treated at start of treatment with alpelisib with any of the following drugs:

     Drugs known to be strong inhibitors or inducers of isoenzyme CYP3A4 including herbal medications, or drugs with a known risk to induce Torsades de Pointes (See Appendix 1, Table 2 for a full list of prohibited medications).

     Note: The patient must have discontinued strong inducers for at least one week and must have discontinued strong inhibitors before the treatment with alpelisib is initiated. Switching to a different medication prior to starting treatment with alpelisib is allowed.
  7. Patient is currently receiving warfarin or other coumarin derived anti-coagulant for treatment, prophylaxis or otherwise. Therapy with heparin, low molecular weight heparin (LMWH), or fondaparinux is allowed.
  8. Patients who have other concurrent severe and/or uncontrolled medical conditions that would, in the Treating Physician's judgment, contraindicate patient participation in the individual patient program (eg. active or uncontrolled severe infection, chronic active hepatitis, immuno-compromised, acute or chronic pancreatitis, uncontrolled high blood pressure, interstitial lung disease, etc.)
  9. Patient has a known history of HIV infection (testing not mandatory) infection
  10. Patient has any of the following cardiac abnormalities:

      a. Symptomatic congestive heart failure i. History of documented congestive heart failure (New York Heart Association functional classification III-IV), documented cardiomyopathy ii. Left Ventricular Ejection Fraction (LVEF) <50% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO) b. Myocardial infarction ≤ 6 months prior to enrolment c. Unstable angina pectoris Acute coronary angioplasty, or stenting), < 3 months prior to screening coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass graft (CABG).

      d. Serious uncontrolled cardiac arrhythmia History or current evidence of clinically significant cardiac arrhythmias, atrial fibrillation and/or conduction abnormality, e.g. congenital long QT syndrome, high-grade/complete AV-blockage: per guidelines.

      e. Symptomatic pericarditis f. QTcF > 480 msec on the screening ECG (using the QTcF formula) currently receiving treatment with medication that has a known risk to prolong the QT interval or inducing Torsades de Pointes, and the treatment cannot be discontinued or switched to a different medication prior to starting treatment with alpelisib.
  11. Patient has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of alpelisib (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
  12. Patient has other prior or concurrent malignancy (except for the following: adequately treated basal cell or squamous cell skin cancer, or other adequately treated in situ cancer, early gastric or GI cancer resected completely by endoscopy procedures or any other cancer from which the patient has been disease free for ≥ 3 years)
  13. Patient has a history of non-compliance to medical regimen or inability to grant consent
  14. Patient who does not apply highly effective contraception during the treatment with alpelisib and through the duration as defined below after the final dose of alpelisib:

      1. Sexually active males should use a condom during intercourse while taking drug and for 4 weeks* after the final dose of alpelisib and should not father a child in this period, but may be recommended to seek advice on conservation of sperm. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid.
      2. Women of child-bearing potential, defined as all female physiologically capable of becoming pregnant, must use highly effective contraception during the IPP and through at least 4 weeks* after the final dose of alpelisib
      3. Highly effective contraception is defined as either:

      i. Total abstinence: When this is in line with the preferred and usual lifestyle of the subject. [Periodic abstinence (e.g., calendar, ovulation, symptothermal, postovulation methods) and withdrawal are not acceptable methods of contraception].

      ii. Female sterilization: have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy or tubal ligation at least six weeks before starting treatment with alpelisib. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment iii. Male partner sterilization (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate). [For female patients participating to this IPP, the vasectomized male partner should be the sole partner for that patient] iv. Use a combination of the following (both a+b):
      1. Placement of an intrauterine device (IUD) or intrauterine system (IUS)
      2. Barrier methods of contraception: Condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository.

      Note: Hormonal contraception methods (e.g. oral, injected, and implanted) are not allowed as alpelisibBYL719 may decrease the effectiveness of hormonal contraceptives.

      * Please consult your local product labels should any concomitant medications be used, as this period may be longer for other potentially genotoxic compounds.

      A female is considered post-menopausal and not of child-bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) at least six weeks ago before the treatment start. For females with therapy-induced amenorrhea, oophorectomy or serial measurements of Follicle-Stimulating Hormone (FSH) and/or estradiol are needed to ensure postmenopausal status.

      NOTE: Ovarian radiation or treatment with a luteinizing hormone-releasing hormone (LHRH) agonist (goserelin acetate or leuprolide acetate) is not permitted for induction of ovarian suppression.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Ian Rabinowitz, MD, Principal Investigator — University of New Mexico Cancer Center
Locations (1):
- University of New Mexico - Cancer Center, Albuquerque, New Mexico, United States

REFERENCES:
- [Derived] Shaheen MF, Tse JY, Sokol ES, Masterson M, Bansal P, Rabinowitz I, Tarleton CA, Dobroff AS, Smith TL, Bocklage TJ, Mannakee BK, Gutenkunst RN, Bischoff J, Ness SA, Riedlinger GM, Groisberg R, Pasqualini R, Ganesan S, Arap W. Genomic landscape of lymphatic malformations: a case series and response to the PI3Kalpha inhibitor alpelisib in an N-of-1 clinical trial. Elife. 2022 Jul 5;11:e74510. doi: 10.7554/eLife.74510. PMID 35787784

DOCUMENTS (1):
  • Study Protocol (2017-01-19): https://cdn.clinicaltrials.gov/large-docs/82/NCT03941782/Prot_000.pdf